CLINICAL TRIAL: NCT06219694
Title: Enhancing Chronic Migraine Preventive Therapy: Laser Acupuncture as an Add-On Treatment for Patients With Unsatisfactory Pharmacological Effect, a Pilot Randomized Controlled Trial
Brief Title: Laser Acupuncture for Chronic Migraine
Acronym: LAFCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CF22082B
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Chronic Migraine
Keywords: Migraine; Chronic Migraine; laser acupuncture; Prevention
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: The patients was divided to sham group or laser acupuncture group. After 1 months treatment, and followed up for > 6 months., the sham group received complementary laser acupuncture for 1 months and followed up for another 3 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were randomized by computer software (Excel 2016 for Windows) and the randomization process was overseen by the Institutional Review Board at Taichung Veterans General Hospital. All the participants and our collaborative case-manager were blinded to treatment types.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture (Experimental): CM patients with unsatisfactory pharmacological effects receive laser acupuncture for 8 sessions that spanned 4 weeks. Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  Interventions: Device: Laser Acupuncture
- Sham treatment (Sham Comparator): CM patients with unsatisfactory pharmacological effects receive sham treatment for 8 sessions that spanned 4 weeks. Sham treatment had no laser output.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Laser Acupuncture — Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  Arms: laser acupuncture
Device: Sham — Sham treatment with no laser output, stimulate the same acupoints as laser acupuncture group as follows: 30 seconds at bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  After > 6 months followed up, the sham group received truely Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3), and followed up for another 3 months.
  Arms: Sham treatment

SUMMARY:
A single-blind randomized controlled trial was conducted from October 2024 to May 2025. Chronic migraine patients were randomly assigned in a 1:1 ratio to receive either Laser acupuncture or sham treatment. The co-primary outcomes were changes in monthly migraine days (MMD) and acute headache medications usage days per month from baseline, and Hospital Anxiety and Depression Scale (HADS), and Beck's Depression Inventory(BDI) evaluation. Evaluations were taken at baseline and each follow-up point.

After >6 months follow up as washing out time, the sham group received complementary laser acupuncture treatment and follow up for another 3 months, compared the Headache related parameters (onset, duration, pain scale, current medication for headache, menstrual cycle).

DETAILED DESCRIPTION:
Headache is one of the most common complaints encountered in medical institution as known as an almost universal human experience. Approximately 65% of headaches are classified as primary, which was a composite of migraine, tension-type headache, trigeminal autonomic cephalalgia and other primary headaches according to the third edition of the International Classification of Headache Disorders (ICHD-3). Primary headaches encompass a heterogeneous group of neurologic disorders and might be bothersome for patients.

It's well established that acupuncture can be considered a treatment option for migraine prevention. The efficacy of laser-acupuncture is similar to acupuncture, and laser-acupuncture is a non-invasive therapeutic approach and safety. It could reduce the risk of hemorrhage, infection and needle phobia. However, the efficacy of laser-acupuncture in primary headache remains inconclusive.

Aims:

We aimed to investigate the efficacy and safety of laser acupuncture (LA) as an add-on preventive therapy on chronic migraine (CM).

Methods In this hospital-based prospective single blind randomized sham-controlled study, patients over 18 years old with primary headache will be randomly divided into two treatment arms including laser-acupuncture and sham-controlled group. The expected laser-acupuncture protocol will be bilateral BL2, GB20, EX-HN5, GB8, LI4, LR3 and midline EX-HN3 in totally eight sessions at the first month. In the sham-laser-acupuncture group, patients will receive eight sessions of laser-acupuncture for free after unblinding. We expected to track patients for at least half year. The diagnosis and classification of headache was evaluated using the ICHD-3 criteria. The severity of headache was evaluated using Migraine Disability Assessment (MIDAS) and headache diary provided by Taiwan Headache Society. The co-primary efficacy end points are change in migraine days per month and variation of MIDAS. The secondary end point is the reducing of the severity of comorbidities including headache related anxiety and depression, and both of the quality of life and sleep.

In addition, patients' characteristics will be investigated as follows:

1. Sociodemographic factors (ethnicity, age, sex, body weight, BMI, blood pressure)
2. Headache related parameters (onset, duration, pain scale, current medication for headache, menstrual cycle)
3. Anxiety, evaluate by Hospital Anxiety and Depression Scale (HADS)
4. Depression, evaluate by Beck's Depression Inventory
5. Quality of life, evaluate by 36-Item Short Form Survey (SF-36)
6. Quality of sleep, evaluate by Pittsburgh Sleep Quality Index (PSQI)
7. Aura of headache
8. Episodic or chronic headache (If patient diagnosed as migraine.)
9. Nausea, vomiting, photophobia, phonophobia (If patient diagnosed as migraine.)

A single-blind randomized controlled trial was conducted from October 2024 to May 2025. CM patients with unsatisfactory pharmacological effects were randomly assigned in a 1:1 ratio to receive either LA or sham treatment over a course of 8 sessions spanning 4 weeks. Evaluations were taken at baseline (12 weeks before randomization), at 4th week (treatment completed), 8th week and 12th week from baseline, and follow up till > 24th week, and the sham group received complementary laser acupuncture treatment and follow up for another 3 months, compared the Headache related parameters (onset, duration, pain scale, current medication for headache, menstrual cycle).

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 20 years old and had CM managed pharmacologically, including preventive and/or acute migraine medications, and in addition, those who had refused preventive agent despite recommendation of the neurologist;
* patients who had unsatisfactory effect of current pharmacological treatments, defined as they self-reported
* patients who had a minimum of one-year history of migraine with or without aura.

Exclusion Criteria:

* patients who had received another LA therapy or traditional acupuncture at baseline
* migraine onset after the age of 50
* cognitive or psychological impairment interfering with the participant's ability to receive LA protocol and describe symptoms
* patients with missing data at baseline or during the follow-up period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
monthly migraine days | 12 weeks, 24 weeks, 36 weeks
  change in monthly migraine days (MMD) from baseline and each follow-up time point
acute headache medications usage days | 12 weeks, 24 weeks, 36 weeks
  change in acute headache medications usage days per month from baseline and each follow-up time point

SECONDARY OUTCOMES:
30% reduction in migraine days | 12 weeks, 24 weeks, 36 weeks
  ≥ 30% reduction in migraine days between baseline and each follow-up time point
headache duration | 12 weeks, 24 weeks, 36 weeks
  changes in the headache duration between baseline and each follow-up time point
headache severity | 12 weeks, 24 weeks, 36 weeks
  changes in the headache severity (based on NRS) between baseline and each follow-up time point
the MIDAS score | 12 weeks
  changes in the MIDAS score between baseline and each follow-up time point
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  change in HADS score between baseline and each follow-up time point
Beck's Depression Inventory | 12 weeks
  change in BDI score between baseline and each follow-up time point

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Chen Liu, M.D, Study Director — Taichung Veterans General Hospital; Ching-Chun Chung, M.D, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Xitun District, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT06219694/Prot_SAP_000.pdf